CLINICAL TRIAL: NCT06204562
Title: Feasibility and Effects of Laughter-imitation Therapy (LIT) in Promoting Mental Wellbeing Among Institutional Older Adults
Brief Title: Feasibility and Effects of Laughter-imitation Therapy (LIT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UW 23-424
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Aging Well

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-month imitated laughter practice (Experimental): The intervention is one-month imitated laughter practice. Each practice session lasts for 3 minutes once a day, giving a total of 21 minutes per week. A brief one-to-one training will be offered and a trained research assistant (RA1). Further in-person demonstration and return demonstration will be conducted until participant is able to demonstrate the Duchenne smile on their own. RA1 will be on-site for two days in the first week and one day in the second week to support the participants.
  Interventions: Behavioral: imitated laughter practice
- waitlist control (Experimental): The waitlist control group will be under usual care for the first 8 weeks. Then, they will start intervention after the 8 week, and receive two additional outcome assessments.
  Interventions: Behavioral: imitated laughter practice

INTERVENTIONS:
Behavioral: imitated laughter practice — To imitate laughter, participants will practice "Duchenne smile", which is reported to associate with positive emotion in people producing it If participants cannot imitate a Duchenne smile, they can hold a chopstick horizontally in their mouth tightly. To help timing the 3-minute and to enhance adherence, an audio recording with joyous music and vocal instruction will be played alongside the practice. Versions with or without laugh voice will be prepared for their preferences. A logbook will be given to each participant to record their practice. To remind participants to practise, a reminder will be made each day through the public announcement system of the respective nursing home, and the audio guide will be played.

SUMMARY:
Background: The mental wellbeing of the institutional population has to be promoted, particularly after the serious hit by the pandemic.

Objectives:

1. To develop a LIT intervention to promote mental wellbeing of institutional older adults
2. To explore the feasibility and acceptability of such intervention;
3. To explore the potential effect of the intervention

Design and subject:

A pilot cluster randomized control trial will be conducted. The target population is institutional older adults. About 30 participants will be recruited from 2 nursing homes. The intervention is one-month imitated laughter practice. Each practice session lasts for 3 minutes once a day, giving a total of 21 minutes per week and the waitlist control group will be under usual care for the first 8 weeks. Then, they will start intervention after the 8 week, and receive two additional outcome assessments. A brief one-to-one training will be offered and a trained research assistant (RA1). Further in-person demonstration and return demonstration will be conducted until participant is able to demonstrate the Duchenne smile on their own. RA1 will be on-site for two days in the first week and one day in the second week to support the participants. At the end of the intervention, qualitative feedback will be collected from purposive sample until data saturation.

Instruments: Chinese version including the World Health Organization Five Well-Being Index (WHO-5), 4-item Subjective Happiness Scale (SHS), Geriatric Depression Scale (GDS), Pittsburgh Sleep Quality Index (PSQI), 5-min Montreal Cognitive Assessment, FRAIL scale, Geriatric Adverse Life Events Scale (GALES).

Main outcome measures: Feasibility and acceptability of laughter-imitation therapy (LIT)

Data analysis: Descriptive statistics will be calculated for participants' characteristics, practice frequency, satisfaction, and health outcomes. Linear mixed-effects models will be used to evaluate health outcomes. Content analysis will be conducted for qualitative feedback.

Expected results: The intervention is expected to be feasible and acceptable to institutional older adults as a means for promoting mental wellbeing, and potential beneficial effects will be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

i. aged ≥65 years, ii. living in institutions for ≥6 months and will continue to live there for ≥6 months, iii. no communication problems, iv. cognitively capable (screened by 5-min Montreal Cognitive Assessment (MoCA) > age-and-education specific cutoff at 7th-percentile).

Exclusion Criteria:

i. facial paralysis or paralysed Zygomaticus major muscle or orbicularis oculi muscle, ii. hearing problem that prevent them from following audio recording, iii. undergoing oxygen therapy that may hinder their practice, iv. those with undiagnosed depression but is detected by screening with Geriatric Depression Scale ≥ 8 (they will be referred to professional service).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Participation rate of laughter-imitation therapy (LIT) | 16 weeks after baseline
  To reflect feasibility, the participation rate, calculated by dividing the number of participants joining the study by the number of participants invited, will be calculated.
Compliance rate of laughter-imitation therapy (LIT) | 16 weeks after baseline
  To calculate the compliance rate, the number of practiced session divided by the number of scheduled session will be estimated. The participants will use a log book (Appendix V) to record their daily practice of self-induced laughter.
Acceptance of laughter-imitation therapy (LIT) | 16 weeks after baseline
  To measure acceptance, level of satisfaction with the intervention will be collected by a single question with five point likert scale.

SECONDARY OUTCOMES:
Change from baseline mental wellbeing at 4 weeks | 4 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). WHO-5 consists of five statements on their mental wellbeing in the past two weeks, using a score from 0 (no time) to 5 (all of the time). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline mental wellbeing at 8 weeks | 8 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). WHO-5 consists of five statements on their mental wellbeing in the past two weeks, using a score from 0 (no time) to 5 (all of the time). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline mental wellbeing at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). WHO-5 consists of five statements on their mental wellbeing in the past two weeks, using a score from 0 (no time) to 5 (all of the time). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline mental wellbeing at 16 weeks | 16 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). WHO-5 consists of five statements on their mental wellbeing in the past two weeks, using a score from 0 (no time) to 5 (all of the time). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline subjective happiness at 4 weeks | 4 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). Participants will respond on a 7-point Likert scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline subjective happiness at 8 weeks | 8 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). Participants will respond on a 7-point Likert scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline subjective happiness at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). Participants will respond on a 7-point Likert scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline subjective happiness at 16 weeks | 16 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). Participants will respond on a 7-point Likert scale. The score is the average of the four items, and ranges from 1 to 7; a higher score indicates a higher happiness level.
Change from baseline depressive symptoms at 4 weeks | 4 weeks after baseline
  Measured by the Chinese version of the Geriatric Depression Scale (GDS). Chinese version of GDS has been validated as a promising screening instrument for depression in Chinese older adult and comprises 15 questions scored in a dichotomous format. Using a cut-off score of 8 is suggested to be the indicator of being depressed.
Change from baseline depressive symptoms at 8 weeks | 8 weeks after baseline
  Measured by the Chinese version of the Geriatric Depression Scale (GDS). Chinese version of GDS has been validated as a promising screening instrument for depression in Chinese older adult and comprises 15 questions scored in a dichotomous format. Using a cut-off score of 8 is suggested to be the indicator of being depressed.
Change from baseline depressive symptoms at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the Geriatric Depression Scale (GDS). Chinese version of GDS has been validated as a promising screening instrument for depression in Chinese older adult and comprises 15 questions scored in a dichotomous format. Using a cut-off score of 8 is suggested to be the indicator of being depressed.
Change from baseline depressive symptoms at 16 weeks | 16 weeks after baseline
  Measured by the Chinese version of the Geriatric Depression Scale (GDS). Chinese version of GDS has been validated as a promising screening instrument for depression in Chinese older adult and comprises 15 questions scored in a dichotomous format. Using a cut-off score of 8 is suggested to be the indicator of being depressed.
Change from baseline sleep quality at 4 weeks | 4 weeks after baseline
  Measured by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). PSQI has been validated as a reliable tool for older adults in Chinese. The 19-item scale covers 7 components and the global PSQI score ranges from 0 to 21 with higher score indicating poorer quality.
Change from baseline sleep quality at 8 weeks | 8 weeks after baseline
  Measured by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). PSQI has been validated as a reliable tool for older adults in Chinese. The 19-item scale covers 7 components and the global PSQI score ranges from 0 to 21 with higher score indicating poorer quality.
Change from baseline sleep quality at 12 weeks | 12 weeks after baseline
  Measured by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). PSQI has been validated as a reliable tool for older adults in Chinese. The 19-item scale covers 7 components and the global PSQI score ranges from 0 to 21 with higher score indicating poorer quality.
Change from baseline sleep quality at 16 weeks | 16 weeks after baseline
  Measured by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). PSQI has been validated as a reliable tool for older adults in Chinese. The 19-item scale covers 7 components and the global PSQI score ranges from 0 to 21 with higher score indicating poorer quality.
Change from baseline pain experience at 4 weeks | 4 weeks after baseline
  Measured by the recall period of one week for pain severity ratings from 0 to 10 with higher score indicating greater severity and methods of pain relief will be evaluated.
Change from baseline pain experience at 8 weeks | 8 weeks after baseline
  Measured by the recall period of one week for pain severity ratings from 0 to 10 with higher score indicating greater severity and methods of pain relief will be evaluated.
Change from baseline pain experience at 12 weeks | 12 weeks after baseline
  Measured by the recall period of one week for pain severity ratings from 0 to 10 with higher score indicating greater severity and methods of pain relief will be evaluated.
Change from baseline pain experience at 16 weeks | 16 weeks after baseline
  Measured by the recall period of one week for pain severity ratings from 0 to 10 with higher score indicating greater severity and methods of pain relief will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Hing Chau, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Community, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No